CLINICAL TRIAL: NCT03650738
Title: A Prospective, One-arm Open Clinical Trial of Apatinib Combined With Albumin Paclitaxel and Carboplatin as a Neoadjuvant Therapy for the Safety and Efficacy of Triple-negative Breast Cancer
Brief Title: This Study Was a Prospective, One-arm Open Phase II Clinical Trial. A Systematic Review of the pCR of Apatinib in Combination With the Albumin Paclitaxel and Carboplatin Regimens for the Neoadjuvant Therapy of Triple-negative Breast Cancer, as Well as the Safety of Treatment
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: The First Affiliated Hospital with Nanjing Medical University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BL2014084
Record Dates: First submitted 2018-08-27; First posted 2018-08-29 (Actual); Last update posted 2018-08-29 (Actual); Status verified 2018-08

CONDITIONS: Systematic Review of the pCR Rate of Apatinib Combined With Albumin Paclitaxel and Carboplatin Regimen for Neoadjuvant Therapy of Triple-negative Breast Cancer
MeSH Terms: interventions — apatinib; Carboplatin

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Study group (Experimental): apatinib 250mg oral d1-21; albumin paclitaxel 260mg/m2 intravenous drip d1; carboplatin AUC=5-6 intravenous drip d1; 21 days for 1 cycle. The treatment regimen was used for a total of 6 cycles, or to PD, or the toxicity was not tolerated.
  Interventions: Drug: Apatinib

INTERVENTIONS:
Drug: Apatinib — Neoadjuvant program: apatinib 250mg oral d1-21; albumin paclitaxel 260mg/m2 intravenous drip d1; carboplatin AUC=5-6 intravenous drip d1; 21 days for 1 cycle. The treatment regimen was used for a total of 6 cycles, or to PD, or the toxicity was not tolerated.
  Other Names: Carboplatin; albumin paclitaxel

SUMMARY:
This study was a prospective, one-arm open phase II clinical trial. A systematic review of the pCR of apatinib in combination with the albumin paclitaxel and carboplatin regimens for the neoadjuvant therapy of triple-negative breast cancer, as well as the safety of treatment, at the same time, relevant exploratory biomarker research is conducted.

DETAILED DESCRIPTION:
Neoadjuvant program: apatinib 250mg oral d1-21; albumin paclitaxel 260mg/m2 intravenous drip d1; carboplatin AUC=5-6 intravenous drip d1; 21 days for 1 cycle. The treatment regimen was used for a total of 6 cycles, or to PD, or the toxicity was not tolerated. If there is still no PD after 6 cycles, the surgical approach is based on the tumor condition and the patient's wishes. If the condition progresses to terminate the treatment regimen, the patient may receive subsequent local or systemic treatment. The follow-up period was followed up to assess safety and effectiveness.

MAIN OBJECTIVE: To systematically evaluate the pCR rate of apatinib combined with albumin paclitaxel and carboplatin regimen for neoadjuvant therapy of triple-negative breast cancer Secondary objective: To evaluate the safety of apatinib combined with albumin paclitaxel and carboplatin in neoadjuvant therapy for triple-negative breast cancer, an exploratory biomarker study

ELIGIBILITY:
Inclusion Criteria:

* 1. The patient volunteers and signs an informed consent form. 2.age ≥18 years old, female; 3.Diagnosed as triple negative breast cancer by histopathology; 4.Did not receive systemic anti-tumor treatment; 5. The clinical stage is stage II-III; 6.There must be at least one measurable lesion (according to RECIST v1.1); 7.Physical condition ECOG PS: 0-1; 8.Expected survival time ≥ 3 months; 9.Laboratory tests meet the following criteria: Bone marrow function: absolute count of blood neutrophils (ANC) ≥1.5×109/L; platelet (PLT)≥100×109/L; hemoglobin (HB)≥90g/L; Liver function: serum total bilirubin (STB), combined bilirubin (CB) ≤ upper limit of normal (ULN) *1.5; alanine aminotransferase (ALT), aspartate aminotransferase (AST) ≤ULN*2.5; Renal function: serum creatinine (Cr) ≤ ULN; endogenous creatinine clearance (Ccr) ≥ 60 ml / min (calculated using the Cockcroft-Gault formula);

Exclusion Criteria:

* 1.Major surgery within 4 weeks prior to enrollment, or surgical wounds have not healed; 2.Embolization and bleeding occurred within 4 weeks before enrollment; 3.Malignant tumors of other histological origins in the past 5 years, except for cured cervical carcinoma in situ and basal cell carcinoma or squamous cell carcinoma; 4.Severe cardiovascular disease, including hypertension (BP≥160/95mmHg) uncontrolled by medical treatment, unstable angina, history of myocardial infarction in the past 6 months, congestive heart failure>NYHA II, severe heart rhythm Abnormalities and pericardial effusions; 5.Severe infection requires intravenous antibiotic, antifungal or antiviral treatment; 6.Suffering from mental illness, poor compliance; 7.Researchers believe that it is not suitable for inclusion.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2018-09-01 (Estimated); Primary Completion 2019-12-30 (Estimated); Study Completion 2019-12-31 (Estimated)

PRIMARY OUTCOMES:
pCR rate | 4 months
  The treatment regimen was used for a total of 6 cycles, or to PD, or the toxicity was not tolerated.

CONTACTS AND LOCATIONS:
Locations (1):
- Jiangsu Provincial Hospital, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No